CLINICAL TRIAL: NCT02591589
Title: The Relationship Between Administered Oxygen Levels and Arterial Partial Oxygen Pressure to Neurocognition in Post-operative Mechanically Ventilated Cardiac Surgical Patients
Brief Title: Intraoperative Oxygen Concentration and Neurocognition After Cardiac Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Shahzad Shaefi, Anesthesiologist, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2014P000398
Record Dates: First submitted 2015-02-13; First posted 2015-10-29 (Estimated); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Hyperoxia; Normoxic; Delirium
Keywords: Hyperoxia; Delirium; Normoxic; t-MoCA
MeSH Terms: conditions — Hyperoxia; Delirium

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normoxic group (Experimental): To standardize key aspects of ventilator support, tidal volume will be set to 6-8ml/kg and PEEP levels will be set to 0-5cm H2O, allowing flexibility for provider preference. For normoxic oxygenation FiO2 will be set at 0.35 (35%) ideally to maintain PaO2 above 70mmHg (or saturations greater than or equal to 92%), and titrated up if need be to prevent potentially injurious hypoxemia (saturations below 92%). During cardiopulmonary bypass, blended air/ oxygen mixture will be titrated to arterial blood gas analysis with maintenance of PaO2 between 100mmHg and 150mmHg.
  Interventions: Other: Normoxic oxygenation
- Hyperoxic group (Active Comparator): To standardize key aspects of ventilator support, tidal volume will be set to 6-8ml/kg and PEEP levels will be set to 0-5cm H2O, allowing flexibility for provider preference. For hyperoxic oxygenation FiO2 will be set at 1.0 (100%) throughout the intraoperative period, including cardiopulmonary bypass.
  Interventions: Other: Hyperoxic oxygenation

INTERVENTIONS:
Other: Normoxic oxygenation — FiO2 set at 0.35 to maintain PaO2 > 70 mmHg or oxygen saturation greater than or equal to 92%.
  Arms: Normoxic group
Other: Hyperoxic oxygenation — FiO2 set at 1.0 throughout the procedure
  Arms: Hyperoxic group

SUMMARY:
This is a randomized, prospective controlled trial in patients undergoing cardiac surgery, specifically on-pump coronary artery bypass grafting, comparing level of administered oxygen and partial pressure of arterial oxygen in the operating room and its impact on a widely-used and validated neurocognitive score, the telephonic Montreal Cognitive Assessment (t-MoCA), throughout the hospital stay and at 1 month, 3 months, and 6 postoperatively. It is hypothesized that cardiac surgical patients who undergo normoxic conditions throughout the intraoperative period will have better neurocognitive function than those with maintenance of hyperoxia.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 65 years and older
* Undergoing elective or urgent on-pump Coronary Artery Bypass Graft (CABG) only

Exclusion Criteria:

* Off-pump or any other procedure in addition to CABG
* Emergent procedure
* One-lung ventilation
* Non-English speaking
* Baseline tMoCA score <10
* Preoperative inotrope use
* Preoperative vasopressor use
* Intra-aortic balloon counterpulsation
* Mechanical circulatory support (Intra-aortic balloon pump (IABP)/ Ventricular assisted devices (VAD)/Extracorporeal membrane oxygenation (ECMO))
* Active cardiac ischemia
* Acute decompensated arrhythmia
* O2 sat < 90% on supplemental oxygen
* Use of continuous vasopressor or inotrope infusion medications
* Significant physician or nurse concern

Cessation Criteria

* Development of significant intraoperative hemodynamic compromise as a result of cardiac surgery
* Oxygen desaturation <90% for > 3 min
* Significant physician or nurse concern

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-07; Primary Completion 2018-01-17 (Actual); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Telephonic-MoCA (t-MoCA) | Change from baseline tMoCA score through 6 months
  t-MoCA will be performed baseline, daily starting POD#1 as well as at 1, 3 and 6 months post-operatively. In previous studies, testing through month 6, has been shown to accurately reflect more longitudinal follow-up. t-MoCA results are on a 22 point scale and will be used as a marker for cognitive function and has been validated. Blinded study staff trained in administering the assessments will collect the data.

SECONDARY OUTCOMES:
Confusion Assessment Method for the ICU | Post-operative day 1 through discharge from hospital (3-5 days on average)
  CAM and CAM-ICU as a marker of delirium post-operatively will be administered and measured at the same time as the t-MoCA. This is a validated test to measure delirium. There is much data to support an increased reduction in cognitive ability in patients exhibiting post-operative delirium.
Days of mechanical ventilation | Post-operative day 1 through discharge from hospital (3-5 days on average)
Length of stay in hospital | Post-operative day 1 through discharge from hospital (3-5 days on average)
Time to extubation | Post-operative day 1 through discharge from hospital
Patient mortality | 30 days and 6 months post-operatively
Biomarkers of oxidative stress, IL-6, IL-8 and others | Intraoperatively at cardiopulmonary bypass (CPB)

CONTACTS AND LOCATIONS:
Overall Officials: Shahzad Shaefi, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kilgannon JH, Jones AE, Parrillo JE, Dellinger RP, Milcarek B, Hunter K, Shapiro NI, Trzeciak S; Emergency Medicine Shock Research Network (EMShockNet) Investigators. Relationship between supranormal oxygen tension and outcome after resuscitation from cardiac arrest. Circulation. 2011 Jun 14;123(23):2717-22. doi: 10.1161/CIRCULATIONAHA.110.001016. Epub 2011 May 23. PMID 21606393
- [Background] Kilgannon JH, Jones AE, Shapiro NI, Angelos MG, Milcarek B, Hunter K, Parrillo JE, Trzeciak S; Emergency Medicine Shock Research Network (EMShockNet) Investigators. Association between arterial hyperoxia following resuscitation from cardiac arrest and in-hospital mortality. JAMA. 2010 Jun 2;303(21):2165-71. doi: 10.1001/jama.2010.707. PMID 20516417
- [Background] Bellomo R, Bailey M, Eastwood GM, Nichol A, Pilcher D, Hart GK, Reade MC, Egi M, Cooper DJ; Study of Oxygen in Critical Care (SOCC) Group. Arterial hyperoxia and in-hospital mortality after resuscitation from cardiac arrest. Crit Care. 2011;15(2):R90. doi: 10.1186/cc10090. Epub 2011 Mar 8. PMID 21385416
- [Background] Trzeciak S, Jones AE, Kilgannon JH, Milcarek B, Hunter K, Shapiro NI, Hollenberg SM, Dellinger P, Parrillo JE. Significance of arterial hypotension after resuscitation from cardiac arrest. Crit Care Med. 2009 Nov;37(11):2895-903; quiz 2904. doi: 10.1097/ccm.0b013e3181b01d8c. PMID 19866506
- [Background] Eastwood G, Bellomo R, Bailey M, Taori G, Pilcher D, Young P, Beasley R. Arterial oxygen tension and mortality in mechanically ventilated patients. Intensive Care Med. 2012 Jan;38(1):91-8. doi: 10.1007/s00134-011-2419-6. Epub 2011 Nov 30. PMID 22127482
- [Background] Pilcher J, Weatherall M, Shirtcliffe P, Bellomo R, Young P, Beasley R. The effect of hyperoxia following cardiac arrest - A systematic review and meta-analysis of animal trials. Resuscitation. 2012 Apr;83(4):417-22. doi: 10.1016/j.resuscitation.2011.12.021. Epub 2012 Jan 5. PMID 22226734
- [Background] Neumar RW. Optimal oxygenation during and after cardiopulmonary resuscitation. Curr Opin Crit Care. 2011 Jun;17(3):236-40. doi: 10.1097/MCC.0b013e3283454c8c. PMID 21415737
- [Background] Janz DR, Hollenbeck RD, Pollock JS, McPherson JA, Rice TW. Hyperoxia is associated with increased mortality in patients treated with mild therapeutic hypothermia after sudden cardiac arrest. Crit Care Med. 2012 Dec;40(12):3135-9. doi: 10.1097/CCM.0b013e3182656976. PMID 22971589
- [Background] O'Driscoll BR, Howard LS. How to assess the dangers of hyperoxemia: methodological issues. Crit Care. 2011;15(3):435; author reply 435. doi: 10.1186/cc10272. Epub 2011 Jun 30. No abstract available. PMID 21722333
- [Background] de Jonge E, Peelen L, Keijzers PJ, Joore H, de Lange D, van der Voort PH, Bosman RJ, de Waal RA, Wesselink R, de Keizer NF. Association between administered oxygen, arterial partial oxygen pressure and mortality in mechanically ventilated intensive care unit patients. Crit Care. 2008;12(6):R156. doi: 10.1186/cc7150. Epub 2008 Dec 10. PMID 19077208
- [Background] Saczynski JS, Marcantonio ER, Quach L, Fong TG, Gross A, Inouye SK, Jones RN. Cognitive trajectories after postoperative delirium. N Engl J Med. 2012 Jul 5;367(1):30-9. doi: 10.1056/NEJMoa1112923. PMID 22762316
- [Background] Laffey JG, Talmor D. Predicting the development of acute respiratory distress syndrome: searching for the "Troponin of ARDS". Am J Respir Crit Care Med. 2013 Apr 1;187(7):671-2. doi: 10.1164/rccm.201301-0168ed. No abstract available. PMID 23540873
- [Background] Newman MF, Kirchner JL, Phillips-Bute B, Gaver V, Grocott H, Jones RH, Mark DB, Reves JG, Blumenthal JA; Neurological Outcome Research Group and the Cardiothoracic Anesthesiology Research Endeavors Investigators. Longitudinal assessment of neurocognitive function after coronary-artery bypass surgery. N Engl J Med. 2001 Feb 8;344(6):395-402. doi: 10.1056/NEJM200102083440601. PMID 11172175
- [Derived] Wiredu K, Mueller A, McKay TB, Behera A, Shaefi S, Akeju O. Sex Differences in the Incidence of Postoperative Delirium after Cardiac Surgery: A Pooled Analyses of Clinical Trials. Anesthesiology. 2023 Oct 1;139(4):540-542. doi: 10.1097/ALN.0000000000004656. No abstract available. PMID 37535937
- [Derived] Shaefi S, Marcantonio ER, Mueller A, Banner-Goodspeed V, Robson SC, Spear K, Otterbein LE, O'Gara BP, Talmor DS, Subramaniam B. Intraoperative oxygen concentration and neurocognition after cardiac surgery: study protocol for a randomized controlled trial. Trials. 2017 Dec 19;18(1):600. doi: 10.1186/s13063-017-2337-1. PMID 29254495